CLINICAL TRIAL: NCT04482153
Title: Prevalence of Non-alcoholic Fatty Liver Disease in Patients With Chronic Kidney Disease in Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed, Principal investigator, Assiut University
Other Study IDs: NAFLD inCKD
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Study of the NAFLD in CKD Patients Using Fibroscan Study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: fibroscan — The Controlled Attenuation Parameter (CAP) can using transient elastography (TE) (Fibroscan®) permits to efficiently separate different grades of severity of steatosis. CAP is based on the properties of ultrasonic signals acquired by the Fibroscan®. It allows to simultaneously measure liver stiffness and CAP in the same liver volume.

SUMMARY:
The aim of our study is:

1. The early detection of NAFLD in CKD patients with different stages (stage I to IV) to avoid progression to liver fibrosis.
2. Evaluation of the relationship between the severity of fatty liver in NAFLD assessed by liver enzymes, biochemical markers, ultrasonography and grades of Fibroscan with CKD staging, eGFR and proteinuria.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is defined as presence of reduced glomerular filtration rate (GFR) < 60 ml/min/ 1.73 m2 and/or evidence of kidney damage (usually indicated by albuminuria or proteinuria) for > 3 months or more irrespective of cause . CKD stages are classified according to the National Kidney Foundation in to five stages according to estimated GFR .

The prevalence of CKD is continuously rising in concert with the rising epidemic of its risk factors including ageing, diabetes, obesity, metabolic syndrome, smoking, and hypertension .

Non-alcoholic fatty liver disease (NAFLD) is one of the most common chronic liver diseases in Western countries. It encompasses a spectrum of conditions with lipid deposition in hepatocytes, ranging from simple steatosis to non-alcoholic steatohepatitis (NASH).

It is defined as fatty liver with inflammation and hepatocelullar injury with or without fibrosis, advanced fibrosis and cirrhosis. Metabolic syndrome with its clinical traits is highly prevalent in patients with NAFLD .

Preliminary data suggest an association between CKD and NAFLD .reported that the prevalence of CKD was significantly higher in patients with NASH compared to patients without NASH.

Moreover, Yassui k documented the presence of moderately decreased eGFR and high frequency of micro-albuminuria in patients with biopsy proven NASH.

The diagnosis of NAFLD/NASH is based on the gold standard of liver biopsy or less reliably on serum liver enzymes or ultrasound imaging. However, liver biopsy has its limitations: apart from being an invasive procedure, connected with serious complications .

Many non-invasive procedures have been intensively applied to detect hepatic steatosis and fibrosis. The Controlled Attenuation Parameter (CAP) can using transient elastography (TE) (Fibroscan®) permits to efficiently separate different grades of severity of steatosis. CAP is based on the properties of ultrasonic signals acquired by the Fibroscan®. It allows to simultaneously measure liver stiffness and CAP in the same liver volume.

The volume used for the measurement by the Fibroscan® is 200 times larger than that of a liver biopsy specimen. Therefore the Fibroscan® is used more and more in clinical practice .

Many biochemical markers can be used for diagnosis of NAFLD such as tissue inhibitor of metalloproteinase 1 (TIMP1), aminoterminal peptide of procollagen III (P3NP) .

Up till now, the relationship between NAFLD and CKD is still poorly understood and under discussed.

ELIGIBILITY:
Inclusion Criteria:

- Eighty CKD patients with different stages (stage I to IV) according to the National Kidney Foundation are recruited from inpatients of renal unit in internal medicine department, Assuit university hospitals. Their GFR will assessed by using CKD EPI equation measured as GFR=166 x(s cr/0.7)-1.209X(0.993)age if female, and GFR=163X(s cr/0.9)-1.209x(0.993)age if male. (Andrews et al 2009).

CKD staging according to GFR by CKD EPI is:

* Stage1 in which GFR>90 mil/min but evidence of kidney damage.
* Stage 2 GFR 60-89 mil/min.
* Stage 3 GFR 30-95 mil/min.
* Stage 4 GFR 15-29 mil/min.
* Stage 5 GFR<15 mil/min. The patients will be enrolled from October 2020 to October 2021.

Exclusion Criteria:

* 1- All Patients with positive hepatitis C virus antibodies. 2- All Patients with positive hepatitis B surface antigen. 3- Congested liver. 4- Drug induced hepatosteatosis (INH, estrogens, methotrexate, steroids, amiodarone, etc.).

  5- Autoimmune liver diseases. 6- Metabolic liver diseases. 7- Alcoholic liver disease. 8- Malignancy. 9- ESRD (stage V) on hemodialysis. 10- Obesity overweight BMI > 30. 11- Metabolic syndrome. 12- Type II DM.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eighty CKD patients with different stages (stage I to IV) according to the National Kidney Foundation are recruited from inpatients of renal unit in internal medicine department, Assuit university hospitals. Their GFR will assessed by using CKD EPI
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The early detection of NAFLD in CKD patients with different stages (stage I to IV) to avoid progression to liver fibrosis. | 1 year
  The early detection of NAFLD in CKD patients with different stages (stage I to IV) to avoid progression to liver fibrosis.
Evaluation of the relationship between the severity of fatty liver in NAFLD assessed by liver enzymes, biochemical markers, ultrasonography and grades of Fibroscan with CKD staging, eGFR and proteinuria. | 1year
  Evaluation of the relationship between the severity of fatty liver in NAFLD assessed by liver enzymes, biochemical markers, ultrasonography and grades of Fibroscan with CKD staging, eGFR and proteinuria.

REFERENCES:
- [Background] Dowman JK, Tomlinson JW, Newsome PN. Systematic review: the diagnosis and staging of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2011 Mar;33(5):525-40. doi: 10.1111/j.1365-2036.2010.04556.x. Epub 2010 Dec 29. PMID 21198708
- [Background] Guha IN, Parkes J, Roderick P, Chattopadhyay D, Cross R, Harris S, Kaye P, Burt AD, Ryder SD, Aithal GP, Day CP, Rosenberg WM. Noninvasive markers of fibrosis in nonalcoholic fatty liver disease: Validating the European Liver Fibrosis Panel and exploring simple markers. Hepatology. 2008 Feb;47(2):455-60. doi: 10.1002/hep.21984. PMID 18038452
- [Background] Hamad AA, Khalil AA, Connolly V, Ahmed MH. Relationship between non-alcoholic fatty liver disease and kidney function: a communication between two organs that needs further exploration. Arab J Gastroenterol. 2012 Dec;13(4):161-5. doi: 10.1016/j.ajg.2012.06.010. Epub 2012 Sep 10. PMID 23432982
- [Background] Ikizler TA. CKD classification: time to move beyond KDOQI. J Am Soc Nephrol. 2009 May;20(5):929-30. doi: 10.1681/ASN.2009030309. Epub 2009 Apr 23. No abstract available. PMID 19389841
- [Background] Kiapidou S, Liava C, Kalogirou M, Akriviadis E, Sinakos E. Chronic kidney disease in patients with non-alcoholic fatty liver disease: What the Hepatologist should know? Ann Hepatol. 2020 Mar-Apr;19(2):134-144. doi: 10.1016/j.aohep.2019.07.013. Epub 2019 Sep 23. PMID 31606352
- [Background] Martinez SM, Crespo G, Navasa M, Forns X. Noninvasive assessment of liver fibrosis. Hepatology. 2011 Jan;53(1):325-35. doi: 10.1002/hep.24013. Epub 2010 Nov 29. PMID 21254180
- [Background] McCullough K, Sharma P, Ali T, Khan I, Smith WC, MacLeod A, Black C. Measuring the population burden of chronic kidney disease: a systematic literature review of the estimated prevalence of impaired kidney function. Nephrol Dial Transplant. 2012 May;27(5):1812-21. doi: 10.1093/ndt/gfr547. Epub 2011 Sep 29. PMID 21965592
- [Background] Shah B, Sucher K, Hollenbeck CB. Comparison of ideal body weight equations and published height-weight tables with body mass index tables for healthy adults in the United States. Nutr Clin Pract. 2006 Jun;21(3):312-9. doi: 10.1177/0115426506021003312. PMID 16772549
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Thomas G, Sehgal AR, Kashyap SR, Srinivas TR, Kirwan JP, Navaneethan SD. Metabolic syndrome and kidney disease: a systematic review and meta-analysis. Clin J Am Soc Nephrol. 2011 Oct;6(10):2364-73. doi: 10.2215/CJN.02180311. Epub 2011 Aug 18. PMID 21852664
- [Background] Yasui K, Sumida Y, Mori Y, Mitsuyoshi H, Minami M, Itoh Y, Kanemasa K, Matsubara H, Okanoue T, Yoshikawa T. Nonalcoholic steatohepatitis and increased risk of chronic kidney disease. Metabolism. 2011 May;60(5):735-9. doi: 10.1016/j.metabol.2010.07.022. Epub 2010 Sep 3. PMID 20817213